CLINICAL TRIAL: NCT02741752
Title: The Influence of Cortical Bone Perforation on Guided Bone Regeneration in Humans: A Randomized Clinical Trial
Brief Title: The Influence of Cortical Bone Perforation on Guided Bone Regeneration in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, seyedamir Danesh Sani, Principal Investigator, postgraduate resident, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 97345
Record Dates: First submitted 2016-04-11; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Alveolar Bone Loss
Keywords: histomorphometry
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Cerebral Decortication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test group (Experimental): decortication group
  Interventions: Procedure: Decortication
- control (No Intervention): without decortication

INTERVENTIONS:
Procedure: Decortication — cortical bone perforation
  Arms: test group

SUMMARY:
The purpose of this randomized clinical trial was to evaluate the effect of cortical bone decortication on the angiogenesis and osteogenesis of augmented ridge by GBR.

DETAILED DESCRIPTION:
Background: The purpose of the current study was to evaluate the effect of cortical bone perforation on angiogenesis and osteogenesis of augmented ridge by guided bone regeneration.

Methods: Fourteen patients (mean age: 52) who were in need of dental implants at areas with osseous defects in the mandible were selected. In the test group (n=7), alveolar cortical bone at the area of regeneration was perforated using a #2 high speed round bur. No decortication of cortical bone was performed in the control group (n=7). Subsequently, defects were augmented by guided bone regeneration using resorbable membrane and bovine bone. After a healing period of 7 months, implant sites were created and trephine cores harvested for histological and histomorphometric analysis of the grafted areas.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were presence of atrophic mandibular ridges with bucco-lingual width ranging between 2-5 mm, as measured on serial sections of a computerized axial tomography (CAT) scan.

Exclusion Criteria:

* Exclusion criteria included patients with diabetes, osteoporosis or other metabolic disorders, smokers, pregnant patients and patients who had any systemic or local factors that would inhibit normal wound healing process.

Ages: 25 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The amount of vital bone formation by histomorphometric analysis after cortical bone perforation | 7 months

IPD SHARING:
Plan to Share IPD: Undecided
AA